CLINICAL TRIAL: NCT03367416
Title: Test of an Organizational Change Model in Dental Care Settings
Brief Title: Organizational Change in Dental Care
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Medical College of Wisconsin (Other); Marquette University (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2017-1247; U56DE027442 (NIH)
Record Dates: First submitted 2017-11-27; First posted 2017-12-08 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Patient No Show
MeSH Terms: conditions — No-Show Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: This study will test the NIATx model, an evidence-based behavioral intervention for implementing organizational change and quality improvement in community based health settings with a high proportion of underserved individuals. The goal of the study will be to use the model to identify and implement organizational changes in dental practices that will improve the no-show rate in underserved populations.
  Interventions: Behavioral: NIATx model

INTERVENTIONS:
Behavioral: NIATx model — The NIATx model engages organizations through a multi-clinic learning collaborative and coaching. NIATx teaches organizations how to implement change by using their own organization as the teaching mechanism. Key components of the model include:
  1. educating executives on how to promote effective process change techniques
  2. training staff teams in the theory and practice of organizational change techniques
  3. training staff to develop and implement a process improvement intervention
  4. implementing a sustainability plan to institutionalize change and avoid reverting to previous methods

SUMMARY:
The proposed research will test the ability of the NIATx Organizational Change Model to improve patient no-show rates as compared to typical training approaches used in dental offices. The purpose of the pilot study is to improve no-show rates and, in the process, test an evidence-based organizational change model that can increase use of evidence-based practices in dental care.

NIATx is not an acronym, it is a proper noun.

DETAILED DESCRIPTION:
For designing the pilot study, it is assumed that the no-show rates in dental clinics will have similar characteristics and response patterns to previous studies.

The preliminary summary data provided by the participating dental clinics, the current average no-show rate is approximately 20%, which would reduce to 10% using the upper limit of the confidence interval from the preliminary data. Based on a simulation study incorporating the above assumptions, with 5 sites each contributing 160 appointments before and after the intervention, the study will have 84% power to detect the hypothesized effect (OR=0.44) at a two-sided 5% significance level. The probability of observing a decrease in no-show rates in at least 4 out of 5 of the clinics is approximately 90%. We expect over 80 appointments per month in each clinic, so the target number of appointments would be expected to be available in 2-3 months.

For the NIATx Fidelity Scale, if an organization has an average score of 2 or higher on the NIATx Fidelity Scale for 8 of the 13 measures that will be considered significant. In a previous study using a similar process, 73% of the organizations that achieved gains of +10%, had 8 measures or more with an average score of 2 or greater, compared to 40% of those who had gains at <10%.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, staff must be:

* 18 or older
* A paid staff member at a dental clinic participating in the study
* Willing to participate in the interviews and share their ideas and experiences
* Involved in an organizational improvement project at a participating clinic
* Be able and willing to provide verbal consent

Exclusion Criteria:

An individual who does not regularly interact with patients in a dental clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community dental clinics that:
  * Serve at least a 50 percent minority population
  * Accept a high number of Medicaid patients
  * Are able to provide de-identified clinic data to the research team
  * Are willing to undertake and support an organizational improvement project to decrease no-show rates
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Analyze clinic data for trends and patterns in patient no-show behaviour. | 7 months
  Data from clinic patient records will be gathered and analyzed to determine the percent of cancelled appointments in a given time period, to detect patterns over time and determine if no-shows are more prevalent with certain populations or procedures.
Staff surveys to test clinic adherence to the components of the NIATx model. | 7 months
  Paper surveys will be used to collect data from clinic staff. Surveys will measure how the clinic conducts organizational change, the degree to which the clinics are using elements of the NIATx model and which proven no-show practices clinics have adopted.
Patient qualitative interviews to assess the patient experience in missing an appointment. | 2 months
  Interviews will be open questions to understand the process from the users point of view. This information will help the study team understand the root causes of patient behaviour and propose model improvements that address these causes.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Molfenter, PhD, Principal Investigator — University of Wisconsin, Madison; Christopher Okunseri, BDS, Principal Investigator — Marquette University
Locations (4):
- United States (4):
  - More Smiles Wisconsin, Madison, Wisconsin
  - Community Dental Clinic North-Marquette School of Dentistry, Milwaukee, Wisconsin
  - Community Dental Clinic South-Marquette School of Dentistry, Milwaukee, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIATx website — https://niatx.net/Home